CLINICAL TRIAL: NCT01805635
Title: Evaluation of the Relationship Between the Parameters of Pulmonary Function (PF) and the Concentration of Fractional Exhaled Nitric Oxide (FeNO) and Clinical Characteristics in Children Being Diagnosed Due to Suspicion of Allergic Diseases
Brief Title: PF and FeNO and Clinical Characteristics in Children Being Diagnosed Due to Suspicion of Allergic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, MDPhDProf, Medical University of Lodz
Other Study IDs: RNN/23/13/KE
Record Dates: First submitted 2013-02-25; First posted 2013-03-06 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Asthma; Allergic Rhinitis; Atopic Dermatitis; Urticaria; Healthy
Keywords: Children; Asthma; Allergic rhinitis; Atopic dermatitis; Urticaria; Healthy
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Dermatitis, Atopic; Urticaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — IgE specific allergen antibodies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children suspected of allergic diseases: Children suspected of allergic diseases No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study is to assess the influence of kind of allergic disease, allergic profile, allergen exposure, treatment method on lung function parameters, fractional exhaled nitric oxide level in children suspected and being diagnosed due to allergic diseases.

DETAILED DESCRIPTION:
The aim of this study is to assess the influence of kind of allergic disease, allergic profile, allergen exposure, treatment method on lung function parameters, fractional exhaled nitric oxide (FeNO) level in children suspected and being diagnosed due to allergic diseases.

Study will be retrospective, conducted in all children diagnosed in the years of 2005-20012 in Laboratory of lung function tests of Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland. The investigators will analyse 5500 male an female children 5-18 year old suspected and being diagnosed due to allergic diseases. In these children nearly 3000 FeNO measurements, 65000 spirometry measurements, 22000 whole-body plethysmography measurements and 48000 occlusion resistance measurements were performed between the years of 2005-2012.

The investigators will retrospectively evaluate following data from medical documentation of patients:

1. FeNO levels.
2. Allergic disease diagnosis.
3. Immunoglobulin E (IgE) specific levels.
4. Treatment (drugs and dosages).
5. Lung function parameters (spirometry, whole-body plethysmography, occlusion resistance, bronchial reversibility test).

ELIGIBILITY:
Inclusion Criteria:

* Children with allergic diseases, healthy children.

Exclusion Criteria:

* Other serious diseases.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with allergic diseases, healthy children.
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Allergic disease diagnosis | 7 years
  Allergic disease diagnosis. The diagnosis and the severity of asthma, allergic rhinitis and atopic dermatitis and other allergic diseases universally established by the doctors (allergologists) according to standard definitions of diseases in the latest guidelines

SECONDARY OUTCOMES:
Lung function (LF) | 7 years
  spirometry, whole-body pletysmography, occlusion resistance, bronchial reversibility test

OTHER OUTCOMES:
Fractional exhaled nitric oxide (FeNO) | 7 years
  Fractional exhaled nitric oxide (Sievers equipment)
Immunoglobulin E (IgE) allergen specific | 7 years
  Immunoglobulin E (IgE) allergen specific (ELISA method)
Treatment of asthma (drugs and dosages) | 7 years
  Treatment of asthma (drugs and dosages last 3 months before measurement of lung function parameters and FeNO)

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Stelmach, MDPhDProf, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland; Tomasz Grzelewski, MDPhD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland

REFERENCES:
- [Derived] Grzelewski T, Stelmach W, Stelmach R, Janas A, Grzelewska A, Witkowski K, Makandjou-Ola E, Majak P, Stelmach I. Spirometry-Adjusted Fraction of Exhaled Nitric Oxide Allows Asthma Diagnosis in Children, Adolescents, and Young Adults. Respir Care. 2016 Feb;61(2):162-72. doi: 10.4187/respcare.04092. Epub 2015 Dec 1. PMID 26628565
- [Derived] Jerzynska J, Janas A, Galica K, Stelmach W, Woicka-Kolejwa K, Stelmach I. Total specific airway resistance vs spirometry in asthma evaluation in children in a large real-life population. Ann Allergy Asthma Immunol. 2015 Oct;115(4):272-6. doi: 10.1016/j.anai.2015.07.002. Epub 2015 Jul 26. PMID 26216360
- [Derived] Grzelewski T, Witkowski K, Makandjou-Ola E, Grzelewska A, Majak P, Jerzynska J, Janas A, Stelmach R, Stelmach W, Stelmach I. Diagnostic value of lung function parameters and FeNO for asthma in schoolchildren in large, real-life population. Pediatr Pulmonol. 2014 Jul;49(7):632-40. doi: 10.1002/ppul.22888. Epub 2013 Sep 9. PMID 24019244